CLINICAL TRIAL: NCT04739436
Title: Evaluation of Unilateral vs Bilateral Hearing Aids for the Treatment of Age-related Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106077; PCORI-HL-2019C1-16059 (Other: PCORI)
Record Dates: First submitted 2021-01-26; First posted 2021-02-04 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bilateral hearing aid fitting group (Other)
  Interventions: Device: Hearing amplification
- Unilateral hearing aid fitting group (Active Comparator)
  Interventions: Device: Hearing amplification

INTERVENTIONS:
Device: Hearing amplification — Bilateral vs. unilateral hearing aids for hearing loss

SUMMARY:
This study aims to evaluate the benefit of bilateral hearing aid use compared to a unilateral hearing aid. Patients with mild to moderate bilateral hearing loss who are considering the purchase of a commercially available hearing aid will be considered for participation. Eligible participants will be randomized to one of the following treatment arms: (1) a bilateral hearing aid fitting group, and (2) a unilateral hearing aid fitting group.

DETAILED DESCRIPTION:
Primary objectives:

1. To compare the hearing-aid benefit of unilateral versus bilateral fittings of commercially-available hearing aids that incorporate a dome coupling (open or closed dome as required by degree of hearing loss, or custom coupling if clinically indicated), which represents the most popular style used for mild to moderate hearing loss.
2. To compare other multi-dimensional outcomes including hearing-related quality of life, hearing aid satisfaction in patient-nominated goals, ecological hearing aid outcomes, and hearing aid use.

Secondary objectives:

1. To compare performance outcomes for unilateral versus bilateral hearing aid fittings
2. To explore the differences in long-term patient reported outcomes for their final hearing aid configuration choice
3. To explore patient experiences in each group (unilateral vs bilateral), and patient preference in regards to their choice of final hearing aid configuration.

This study is being conducted at Duke and Vanderbilt Medical Centers, with Duke functioning as the main coordinating center. Study participants will pay out of pocket for the hearing aid(s), but will be able to extend the hearing aid fitting trial period from 60 days (standard of care) to 180 days (6 months). Participants will be given the opportunity to change their hearing aid configuration and/or return their hearing aid(s) for a refund after 3 months, and again at the end of the 6 month study period.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years of age
* Ability to read and understand English
* Mild to moderate sensorineural hearing loss (defined by a pure-tone average at 500, 1000, and 2000 Hz of <55 dB HL in each ear, and the 3000 Hz and 4000 Hz threshold <80 in each ear), based on a hearing test obtained within the last 6 months by a licensed audiologist.
* Symmetrical hearing loss defined by <20 dB difference between the pure-tone average of 500, 1000, and 2000 Hz between ears)
* Interested in purchasing hearing aids, but is open minded about trying one or two hearing aids
* No prior hearing aid use longer than 3 months (as documented via self-report)
* Adequate literacy to complete questionnaires
* Willing to purchase study-specific hearing aid(s)
* Access to a smart phone and the internet

Exclusion Criteria:

* Concerns for middle ear pathology (e.g., air bone gap of >15 dB at 2 consecutive octave frequencies in either ear)
* Concerns for retrocochlear pathology by audiologist (e.g unilateral tinnitus or ear fullness, referral to ENT/Auditory Brainstem Response testing to r/o acoustic neuroma)
* Severe tinnitus as the reason for seeking amplification
* Co-morbid condition that would interfere with study (e.g., dementia, blindness, neurologic pathology)
* History of fluctuating hearing loss

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Smith, AuD,PhD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Open access to de-identified, coded IPD will be made available via Duke's Research Data Repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were found to be ineligible after randomization, so they are excluded from the number who started the study.
Period: Overall Study
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Started | 140 | 136
Completed | 114 | 107
Not Completed | 26 | 29
Not completed — Lost to Follow-up | 21 | 23
Not completed — Withdrawal by Subject | 4 | 6
Not completed — not randomized properly | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant that started the study in the Bilateral hearing aid fitting group was subsequently excluded from analysis due to not being properly randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group | Total
Number analyzed (Participants) | 139 | 136 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.49 (7.87) | 70.34 (7.87) | 70.92 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 67 | 148
  Male | 58 | 69 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 132 | 130 | 262
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 134 | 127 | 261
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 139 | 136 | 275

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing Aid Benefit as Measured by Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The APHAB score ranges from 1 to 99. The change in APHAB score was calculated as the difference between scores at 3 months and baseline, so the range of possible values for the change score is -98 to 98. A lower APHAB score indicates a better benefit; a negative change score indicates greater benefit at 3 months than at baseline.
Time Frame: Baseline, 3 months
Population: The APHAB score could not be obtained for 18 individuals (5 in the bilateral group, 13 in the unilateral group); 16 due to missed 3-month follow-up visit; 2 individuals did not complete the APHAB at the 3 month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 134 | 123
score on a scale | -19.74 (15.18) | -14.41 (13.02)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; A linear regression model was fit with outcome change in APHAB score between 3 months and baseline, predictor hearing aid fitting group (reference=bilateral), and covariate clinical site; Test type: Superiority; p = 0.003, Regression, Linear — Multiple comparisons were not conducted, so no adjustment of the p-value was necessary; Slope = 5.29, 95% CI 2-sided [1.80 to 8.79]

2. Secondary Outcome: Hearing Aid Benefit, as Measured by the Measured by Glasgow Hearing Aid Benefit Profile (GHABP)
Description: The GHABP has a categorical response scale with values of 1-5 for each item (4 pre-defined listening situations and up to 4 patient-nominated listening situations). Responses are converted to a 0-100 scale. Higher post-intervention responses are indicative of more benefit for all questions except for "In this situation, with your hearing aid, how much difficulty do you now have?" where lower scores are better.
Time Frame: 3 months
Population: Outcome measure data missing for 25 individuals at 3 months (9 from bilateral group, 16 from unilateral group). 16 individuals missed the 3-month visit, 8 individuals did not complete the GHABP at the 3-month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: average scores on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 130 | 120
average scores on a scale
  In this situation, what proportion of the time do you wear your hearing aid? | 87.61 (19.30) | 88.25 (21.09)
  In this situation, how much does your hearing aid help you? | 62.64 (23.32) | 59.08 (22.29)
  In this situation, with your hearing aid, how much difficulty do you now have? | 15.56 (12.38) | 19.91 (12.78)
  For this situation, how satisfied are you with your hearing aid? | 70.63 (21.38) | 66.46 (20.58)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the GHABP question means between the groups at 3 months for the question: In this situation, what proportion of the time do you wear your hearing aid?; Test type: Superiority; p = 0.584, Kruskal-Wallis — No adjustments for multiple comparisons were done
Statistical Analysis 2: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the GHABP question means between the groups at 3 months for the question: In this situation, how much does your hearing aid help you?; Test type: Superiority; p = 0.233, Kruskal-Wallis
Statistical Analysis 3: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the GHABP question means between the groups at 3 months for the question: In this situation, with your hearing aid, how much difficulty do you now have?; Test type: Superiority; p = 0.010, Kruskal-Wallis
Statistical Analysis 4: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the GHABP question means between the groups at 3 months for the question: For this situation, how satisfied are you with your hearing aid?; Test type: Superiority; p = 0.129, Kruskal-Wallis

3. Secondary Outcome: Change in Hearing Aid Benefit as Measured by Bamford-Kowal-Bench Speech in Noise (BKB SIN) Test
Description: Speech and noise collocated and the speech reception threshold (SRT) for 50% performance will be calculated (in dB speech-to-noise ratio S/N).
Time Frame: Baseline, 3 months
Population: The BKB SIN test was missing for 17 individuals at 3 months (6 from bilateral group, 11 from unilateral group) 16 due to missed 3- month follow-up visit, 1 individual did not have the BKB SIN test during the 3-month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 133 | 125
dB | -1.51 (3.57) | -1.37 (3.31)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the change from baseline to 3 months in the co-located BKB SIN test scores between the groups; Test type: Superiority; p = 0.946, Kruskal-Wallis; No adjustments for multiple comparisons were done

4. Secondary Outcome: Change in Hearing Aid Benefit as Measured by the Abbreviated Word Auditory Recognition and Recall Measure (WARRM)
Description: The WARRM provides a word-recognition score and a recall score using 20 audio-recorded monosyllabic words distributed across set sizes of 2, 3, 4, 5, and 6 words. the WARRM is reported as percent correct, with higher scores indicating better performance.
Time Frame: Baseline, 3 months
Population: Data was missing from 16 individuals at 3 months (6 from bilateral group, 10 from unilateral group) due to missed 3-month f/u visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: percent correct responses
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 133 | 126
percent correct responses
  Word-recognition percent correct | 15.56 (19.59) | 14.48 (19.12)
  Recall score percent correct | 3.01 (13.48) | 4.72 (14.32)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypotheses are there are no differences in the change from baseline to 3 months in WARRM recognition scores between the groups; Test type: Superiority; p = 0.490, Kruskal-Wallis; No adjustments for multiple comparisons were done
Statistical Analysis 2: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypotheses are there are no differences in the change from baseline to 3 months in WARRM recall scores between the groups; Test type: Superiority; p = 0.323, t-test, 2 sided — No adjustments for multiple comparisons were done

5. Secondary Outcome: Hearing Aid Satisfaction as Measured by Satisfaction With Amplification in Daily Life (SADL) Survey
Description: The SADL is a 15- item questionnaire, 7-item response scale in 1-unit steps, 1 (poorest) to 7 (highest) for each item (reversed for items 2, 4, 7, 13).; A global score is used, which is the mean of scores for all items (excluding questions 11 and 14, if applicable). Higher scores indicate higher satisfaction .
Time Frame: 3 months , 6 months
Population: Data is missing for 18 individuals at 3 months (5 from bilateral group, 13 from unilateral group) 16 due to missed 3 month visit, 2 did not complete the SADL survey during the 3 month visit; and 60 individuals at 6 months (26 from bilateral group, 34 from unilateral group) 54 due to missed 6 month visit, 6 individuals did not complete the SADL at the 6 month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 134 | 123
score on a scale
  3 months | 5.71 (0.75) | 5.7 (0.68)
  6 months: number analyzed (Participants) | 113 | 102
  6 months | 5.63 (0.81) | 5.64 (0.70)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the SADL scores between the groups at 3 months; Test type: Superiority; p = 0.933, t-test, 2 sided — No adjustments for multiple comparisons were done
Statistical Analysis 2: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the SADL scores between the groups at 6 months; Test type: Superiority; p = 0.929, t-test, 2 sided — No adjustments for multiple comparisons were done

6. Secondary Outcome: Change in Hearing Related Quality Life as Measured by Hearing Handicap Inventory for Elderly (HHIE) Survey Completion
Description: The Hearing Handicap Inventory for Elderly (HHIE) survey is a 25 -item questionnaire on a response scale of "yes (4 points), sometimes (2 points) or no (0 points)". Higher score indicates more hearing handicap. Total range of scores at a given timepoint is 0 to 100.
Time Frame: Baseline, 3 months, 6 months
Population: Data is missing for 19 individuals at 3 months (6 from bilateral group, 13 from unilateral group) 16 due to missed 3 month visit, 3 individuals did not complete the HHIE at the 3 month visit; and 68 individuals at 6 months (30 from bilateral group, 38 from unilateral group) 54 due to missed 3 month visit, 14 individuals did not complete the HHIE at the 6 month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: difference in scores on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 133 | 123
difference in scores on a scale
  Baseline to 3 months | -16.89 (15.71) | -14.7 (14.33)
  Baseline to 6 months: number analyzed (Participants) | 109 | 98
  Baseline to 6 months | -19.14 (17.95) | -15.22 (14.77)

7. Secondary Outcome: Change in Complex Ecological Listening as Measured by the Speech Spatial Qualities (SSQ) Survey
Description: The SSQ is a 49-item questionnaire using a response scale ranging from 0 to 10. Higher scores are better.
Time Frame: Baseline, 3 months, 6 months
Population: Outcome measure is missing for 21 individuals at 3 months (7 from bilateral group, 14 from unilateral group) and 72 individuals at 6 months (32 from bilateral group, 40 from unilateral group). Due to missed 3 and 6-month visits, or missing/incomplete SSQ questionnaires from those visits. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: difference in overall scores on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 132 | 122
difference in overall scores on a scale
  Baseline to 3 months | 0.96 (1.27) | 0.58 (1.21)
  Baseline to 6 months: number analyzed (Participants) | 107 | 96
  Baseline to 6 months | 0.83 (1.27) | 0.85 (1.21)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the change from baseline to 3 months in SSQ scores between the groups; Test type: Superiority; p = 0.015, t-test, 2 sided
Statistical Analysis 2: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the change from baseline to 6 months in SSQ scores between the groups; Test type: Superiority; p = 0.886, t-test, 2 sided; No adjustments for multiple comparisons were done

8. Secondary Outcome: Hours of Hearing Aid Use
Description: Average number of hours hearing aid worn, measured by automated data log extracted from hearing aid
Time Frame: 3 months
Population: Hours of hearing aid use in the right ear is missing for 73 individuals (7 from bilateral group, 66 from unilateral group), and left ear use is missing for 93 individuals (9 from bilateral group, 84 from unilateral group). 16 individuals did not complete the 3- month visit; Data was not collected during the 3- month visit for the other individuals. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 132 | 70
hours per day
  Right ear | 10.09 (3.84) | 10.87 (3.36)
  Left ear: number analyzed (Participants) | 130 | 52
  Left ear | 10.01 (3.84) | 10.35 (4.15)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the number of hours of hearing aid use between the groups in the right ear; Test type: Superiority; p = 0.137, t-test, 2 sided; No adjustments for multiple comparisons were done
Statistical Analysis 2: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the number of hours of hearing aid use between the groups in the left ear; Test type: Superiority; p = 0.612, t-test, 2 sided; No adjustments for multiple comparisons were done

9. Secondary Outcome: Hearing Aid Expectations as Measured by the Expected Consequences of Hearing Aid Ownership (ECHO) Survey
Description: The ECHO survey is 15 questions, a 7-item response scale is used in 1-unit steps, 1 (poorest) to 7 (highest) for each item (reversed for items 2, 4, 7, 13). A global score is used, which is the mean of the scores for all items (excluding question 11, if applicable). Higher scores are better (higher expectations).
Time Frame: Baseline
Population: Outcome measure is missing for 18 individuals at 3 months (5 from bilateral group, 13 from unilateral group) due to missing data and/or missed 3-month visits; and 62 individuals at 6 months (27 from bilateral group, 35 from unilateral group), due to missing data and/or missed 6-month visits. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 139 | 136
scores on a scale | 5.01 (0.64) | 5.05 (0.62)

10. Secondary Outcome: Global Hearing Aid Outcomes as Measured by the International Outcome Inventory for Hearing Aids (IOI_HA) Survey
Description: The IOI_HA total score (ranging from 7 to 35) is calculated by summing the response across the 7 item questionnaire. Choices range from the poorest outcome (1 point) to the best outcome (5 points). Higher scores indicate better outcomes.
Time Frame: 3 months, 6 months
Population: Outcome measure is missing for 18 individuals at 3 months (5 from bilateral group, 13 from unilateral group) and 62 individuals at 6 months (27 from bilateral group, 35 from unilateral group). One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 134 | 123
score on a scale
  3 months | 29.81 (3.64) | 29.06 (3.8)
  6 months: number analyzed (Participants) | 112 | 101
  6 months | 29.88 (3.66) | 29.89 (3.56)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the IOI-HA total score between the groups at 3 months; Test type: Superiority; p = 0.108, t-test, 2 sided; No adjustments for multiple comparisons were done
Statistical Analysis 2: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the IOI-HA total score between the groups at 6 months; Test type: Superiority; p = 0.988, t-test, 2 sided — No adjustments for multiple comparisons were done

11. Secondary Outcome: Experience With Hearing Aid Assignment as Measured by a Self-reported Questionnaire
Description: Participants answered the question "How likely are you to recommend assignment to a friend or family member in need of hearing aids" on a 10-point scale (1=not at all likely, 10=very likely/full recommendation)
Time Frame: 3 months
Population: Outcome measure is missing for 30 individuals at 3 months (12 from bilateral group, 18 from unilateral group), due to missing data and/or missed 3-month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 127 | 118
Participants
  Answer 1-6 | 11 | 28
  Answer 7-8 | 24 | 37
  Answer 9-10 | 92 | 53

12. Secondary Outcome: Number of Participants in Each Arm That Chose 0, 1, or 2 Hearing Aids
Description: Measured by participant's final choice of 0, 1, or 2 hearing aids
Time Frame: 3 months
Population: Missing choice at 3 months for 15 individuals (5 from bilateral group, 10 from unilateral group) due to missed 3-month visits. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 134 | 126
Participants
  Chose 0 hearing aids | 1 | 1
  Chose 1 hearing aid | 26 | 48
  Chose 2 hearing aids | 107 | 77

13. Secondary Outcome: Change in Hearing Aid Benefit as Measured by Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The APHAB score ranges from 1 to 99. The change in APHAB score was calculated as the difference between scores at 6 months and baseline, so the range of possible values for the change score is -98 to 98. A lower APHAB score indicates a better benefit; a negative change score indicates greater benefit at 6 months than at baseline.
Time Frame: Baseline, 6 months
Population: Missing data from 54 individuals (25 from bilateral group, 29 from unilateral group) due to missing data and/or missed 6-month visit. One participant from the Bilateral hearing aid fitting group was excluded from the analysis due to not being randomized properly.
Measure: Mean (Standard Deviation); unit: difference of scores on a scale
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
Number analyzed (Participants) | 114 | 107
difference of scores on a scale | -17.76 (14.32) | -15.7 (12.97)
Statistical Analysis 1: Comparison: Bilateral Hearing Aid Fitting Group vs Unilateral Hearing Aid Fitting Group; The null hypothesis is there is no difference in the change in APHAB score from baseline to 6 months between the groups; Test type: Superiority; p = 0.264, t-test, 2 sided; No adjustments for multiple comparisons were done

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Bilateral Hearing Aid Fitting Group | Unilateral Hearing Aid Fitting Group
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/136
Other Adverse Events (participants affected / at risk) | 0/140 | 0/136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT04739436/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04739436/SAP_001.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04739436/ICF_002.pdf